CLINICAL TRIAL: NCT01675648
Title: A Double-blind Randomised Controlled Clinical Trial of Lofexidine Versus Diazepam in the Management of the Opioid Withdrawal Syndrome During Inpatient Detoxification in Singapore
Brief Title: Lofexidine for Inpatient Opiate Detox in Singapore
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Guo Song, Consultant, Head of Research, NAMS IMH, Institute of Mental Health, Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lofex00428
Record Dates: First submitted 2012-08-16; First posted 2012-08-30 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Opiate Dependent Patients Who Are Undergoing Inpatient Detoxification in Singapore
Keywords: Opiate dependent; inpatient detoxification
MeSH Terms: interventions — lofexidine; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lofexidine & Diazepam Placebo (Experimental): Initial Lofexidine dosage starts from 0.8mg per day, it will be gradually increased by increments of 0.4 to 0.8mg per day up to a maximum of 2.2mg daily. After 3 peak dose days, the dosage will be gradually decreased by 0.2 to 0.6mg per day till to 0.2mg of the last lofexidine dosage in Day 10.
  The Diazepam placebo will be administrated to the patients with the same frequency, time and number tablets of diazepam in the active comparator arm.
  Interventions: Drug: Lofexidine; Drug: Placebo for Diazepam
- Diazepam & Lofexidine Placebo (Active Comparator): The initial dosage of Diazepam is 10 mg per day on Day 1&2, the dosage will be increased to 15 mg per day on Day 3&4, subsequently decreased to 10mg per day on Day 5, 5mg per day on Day 6&7, 2mg per day on Day 8&9&10.
  The Lofexidine placebo will be administrated to the patients with the same frequency, time and number tablets of lofexidine in the experimental arm.
  Interventions: Drug: Diazepam; Drug: Placebo for Lofexidine

INTERVENTIONS:
Drug: Lofexidine
  Other Names: BritLofex 0.2mg
  Arms: Lofexidine & Diazepam Placebo
Drug: Diazepam
  Other Names: Apo-Diazepam 5mg and 2mg
  Arms: Diazepam & Lofexidine Placebo
Drug: Placebo for Lofexidine
  Arms: Diazepam & Lofexidine Placebo
Drug: Placebo for Diazepam
  Arms: Lofexidine & Diazepam Placebo

SUMMARY:
In Singapore, opiate substitution medication e.g. methadone is only licensed for use with specific population. The standard treatment is one week of detoxification assisted with diazepam and symptomatic treatment followed by one week of rehabilitation. However, diazepam is highly addictive and widely abused among heroin users and pharmacologically, does not reduce the physical and psychological craving for opioids which can trigger relapse. Many opiate patients undergoing inpatient detoxification leave prematurely (i.e. PID: patient initiated discharge) because of the severity of unpleasant withdrawal symptoms. The purpose of the study is to establish an alternative medication to reduce opiate withdrawal symptoms for use in Singapore by evaluating the clinical efficacy of Lofexidine versus Diazepam in the management of the opiate withdrawal syndrome during inpatient detoxification.

DETAILED DESCRIPTION:
Study Design: This is a randomized, double-blind (double-dummy design) phase IV clinical trial. Patients will be receiving 10 days of Lofexidine plus Diazepam placebo or Diazepam plus Lofexidine placebo. All the patients are expected to complete the 2-weeks inpatient detoxification programme at the NAMS ward. Up to 122 patients (61 in each randomized arm) will be enrolled into the study to ensure that at least 43 patients in each arm complete Day 4 of study treatment programme.

Efficacy Assessments: The primary efficacy outcome measure will be the Objective Opiate Withdrawal Scale (OOWS) scores (range = 0-13) on Day 3 and Day 4 of the treatment phase. The second efficacy outcome measure will be the Short Opiate Withdrawal Scale (SOWS), Opiate Craving visual analogue scale and Pupil size on Day 3 and Day 4, time to dropout (length of stay on the ward) and emotional/psychological symptoms measured every 3 days. Our expected study outcomes are as following:

* Significantly lower mean scores on the Objective Opiate Withdrawal Scale (OOWS) on day 3 and 4 of detox among patients in the lofexidine arm relative to those in the benzodiazepine arm
* Significantly lower mean scores on the Subjective experience of opiate withdrawal scale (SOWS)on day 3 and 4 of detox among patients in the lofexidine arm relative to those in the benzodiazepine arm
* Significantly larger pupil size on day 3 and 4 of detox among patients in the lofexidine arm relative to those in the benzodiazepine arm
* Significantly lower mean craving score on the Visual Analogue Scale on day 3 and 4 of detox among patients in the lofexidine arm relative to those in the benzodiazepine arm
* Significantly longer stay (days) on the ward among patients in the lofexidine arm relative to those in the benzodiazepine arm
* Significantly lower anxiety and depression score on the MAP among patients in the lofexidine arm relative to those in the benzodiazepine arm

Safety Assessment and Monitoring: After signing the informed consent, the subject will undergo screening assessments to determine eligibility for study enrollment; the screen tests include FBC, LFT, Renal function and 12-lead ECG, and urine pregnancy test if female. A complete physical examination will be performed on the first day of screening. From Day 1 till discharge, Vital Signs (e.g. pulse rate, body temperature, blood pressure and respiratory rate) will be closely monitored by the study nurses at the ward, i.e. immediately prior to each lofexidine dose and in addition, 2 hours after the first dose of each dosing day. Should patients show signs of hypotension, the nurse will inform the investigators and they will determine whether or not it is necessary to terminate the patients' participation in the trial. Patients will be required to repeat a 12-lead ECG test when they complete the study or if they drop out of the study. If there is any significant finding from the repeat ECG, it will be followed through by the investigators until resolved. All the adverse events will be documented and followed through until resolved during the study period. The Regular Study Safety Reports inclusive of patients' recruitment, AE/SAE will be generated periodically and sent to an Independent Date & Safety Monitoring Committee (DSMC) for review, the DSMC comprise addiction medicine experts from outside of IMH. Individual patients or the entire study will be discontinued if there is any major safety finding.

Sample Size and Statistical methods: The estimate of 122 subjects (61 per group) for the sample size is based on the following assumptions - mean (SE) OOWS scores on day 4 of 2.4 (0.4000) and 3.9 (2.7713) for the lofexidine and diazepam groups respectively (which implies an expected absolute treatment effect of 1.5), a power of 80%, and allowing for 30% of the patients dropping out before their evaluation on day 4. Thirty percent dropout implies that 86 subjects (43 per group) are required to evaluate the benefit of lofexidine over diazepam. The primary efficacy analysis will be done using the ITT dataset and the safety profile will be described using the safety dataset. All analysis will be conducted by independent statisticians (SCRI).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the DSM-IV criteria for a diagnosis of opiate dependence (as diagnosed by a NAMS psychiatrist).
2. Individuals are voluntarily undergoing inpatient opiate withdrawal treatment at the National Addictions Management Service (NAMS).
3. Agreeable to participating in the clinical trial and will provide written consent.
4. Males or females who are between the ages of 21-55 years. The lower limit of 21 years is in place because of lack of data on younger populations. The upper limit is set at 55 years as the likelihood of having co-morbid physical health problems is greater.
5. Individuals who have a positive urine screen for the presence of opiates (routinely given on first visit to outpatient clinic).

Exclusion Criteria:

1. Are investigator site personnel directly affiliated with this study and their immediate families, immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
2. Are currently enrolled in, or discontinued within the last 30 days from another clinical trial or medical research judged not to be scientifically or medically compatible with this study.
3. A history of allergy/sensitivity to clonidine, lofexidine, imidazole derivatives (e.g. clotrimazole, antifungal) or alpha-2-adrenergic medications.
4. Co-dependency on alcohol, benzodiazepines or any other drug that would require detoxification.
5. A history of major physical illness (cardiovascular disease, cerebrovascular disease, renal impairment, liver disease, epilepsy, symptomatic HIV, Hepatitis B and/or C).
6. Patients with major psychiatric illness (e.g. psychotic disorders, major depression).
7. Patients prescribed analgesic*(*: Opioid analgesic and similar narcotic analgesics), antihypertensive, antiarrhythmic, or antiretroviral medication.
8. Baseline BP > 140/90 mmHg or < 85/55mmHg, and/or baseline PR <55beats/min.
9. Significant abnormal finding from blood tests (FBC, LFT, Renal function) and ECG during screening.
10. Pregnant or breast feeding.
11. Patients are receiving and not willing to stop the drugs which may cause prolong QT interval and hypotension while using concomitant with Lofexidine, e.g. thioridazine, chlorpromazine, tricyclic antidepressants.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To evaluate differences in OOWS (Objective Opiate Withdrawal Scale) | on day 3 and day 4 during inpatient dotex

SECONDARY OUTCOMES:
To evaluate differences in SOWS (Short Opiate Withdrawal Scale) | on day 3 and day 4 during inpatient detox
To evaluate differences in pupil sizes | on days 3 and 4 of inpatient detox
To evaluate differences in craving on the Visual Analogue Scale | on days 3 and 4 of inpatient detox
To evaluate differences in time to drop-out (length of stay on the ward) | time to drop-out
To evaluate differences in emotional/psychological symptoms | every 3 days

OTHER OUTCOMES:
To evaluate the safety of Lofexidine with opiate dependent patients undergoing inpatient detoxification in Singapore | during 14 days of inpatient detox
  Drop of blood pressure and low pulse rate will be our main safety outcome measures among all the adverse events in both the groups; it will be reported in tabular form.

CONTACTS AND LOCATIONS:
Overall Officials: Song Guo, Ph.D, Principal Investigator — NAMS IMH Singapore
Locations (1):
- National Addictions Management Service, Institute of Mental Health, Singapore, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Guo S, Manning V, Yang Y, Koh PK, Chan E, de Souza NN, Assam PN, Sultana R, Wijesinghe R, Pangjaya J, Kandasami G, Cheok C, Lee KM, Wong KE. Lofexidine versus diazepam for the treatment of opioid withdrawal syndrome: A double-blind randomized clinical trial in Singapore. J Subst Abuse Treat. 2018 Aug;91:1-11. doi: 10.1016/j.jsat.2018.04.012. Epub 2018 Apr 25. PMID 29910009